CLINICAL TRIAL: NCT00936858
Title: A Phase II Trial Using RAD001 for Patients With Radioiodine Refractory Thyroid Cancer
Brief Title: RAD001 for Patients With Radioiodine Refractory Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Massachusetts General Hospital (Other); M.D. Anderson Cancer Center (Other); MOUNT SINAI HOSPITAL (Other); Novartis (Industry)
Responsible Party: Principal Investigator, Glenn J. Hanna, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-049
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Results first posted 2021-09-28 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Thyroid Cancer
Keywords: radioiodine refractory thyroid cancer; RAD001
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm A (Experimental): RAD001 will be administered orally as once daily dose of 10 mg (one 10mg tablet or two 5mg tablets) continuously from study day 1 until progression of disease or unacceptable toxicity.
  Interventions: Drug: RAD001

INTERVENTIONS:
Drug: RAD001
  Other Names: Afinitor (everolimus)

SUMMARY:
Since thyroid cancer becomes refractory to radioactive iodine, treatment options are very limited. Tyrosine kinase inhibitors such as sorafenib have recently shown promise. This trial seeks to expand treatment options for this disease with a new, oral drug called RAD001. It is an inhibitor of the mTOR pathway and has shown activity in neuroendocrine cancers of the gastrointestinal tract and has been approved for the treatment of metastatic renal cell cancer.

DETAILED DESCRIPTION:
* RAD001 will be taken once a day in the morning starting on Day 1 and continue until the participant is no longer participating in the study treatment.
* A history and physical exam will be performed the first day of the study and then once a month. Blood tests including coagulation studies, and thyroid studies will be performed monthly. A urine sample will need to be provided on the first day of treatment and then every 2 months. Imaging consisting of a CT or MRI of the neck, chest and abdomen will be done every 8 weeks after starting RAD001.
* Participants will remain on this research study for up to 24 months. However, if the participants doctor feels that they are benefiting from the study drug and they do not have severe side effects, they may be given the option to continue taking RAD001.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced or metastatic thyroid cancer, excluding thyroid lymphomas not amenable to or refractory to surgical resection, external beam radiotherapy, radioiodine or other local therapies.
* Prior therapy with chemotherapy and targeted therapies except for mTor inhibitors is allowed.
* Medullary thyroid cancer with documented evidence of disease progression by modified RECIST within 6 months before study day 1 or symptomatic disease at the time of screening in the absence of documented disease progression.
* Differentiated thyroid cancer with documented evidence of disease progression by modified RECIST within 6 months before study day 1.
* Anaplastic thyroid cancer with disease progression with documented disease progression by modified RECIST within 6 months of study day 1.
* Patients must have at least one measurable site of disease according to RECIST criteria that has not previously irradiated. If the patient has has previous radiation to the marker lesion(s), there must be evidence of progression since radiation.
* 18 years of age or older
* WHO performance status 2 or less
* Adequate bone marrow, liver, and renal function
* Fasting serum cholesterol 300mg/dL or less OR 7.75 mmol/L or less AND fasting triglycerides 2.5x ULN or less

Exclusion Criteria:

* Patients receiving anticancer therapies within last 2 weeks or who have received radiation therapy within 3 weeks of study day 1
* Prior therapy with mTOR inhibitors
* Patients who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery or patients that may require major surgery during the course of the study
* Prior treatment with any investigational drug within the preceding 3 weeks
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent. Topical or inhaled corticosteroids are allowed.
* Patients should not receive immunization with attenuated live vaccines within 2 weeks of study entry or during study period
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
* Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study
* A known history of HIV seropositivity
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001
* Patients with an active, bleeding diathesis
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods
* Patients who have received prior treatment wih an mTOR inhibitor
* Patients with a known hypersensitivity to RAD001 or other rapamycins or to its excipients
* History of noncompliance to medical regimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Hanna, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mt. Sinai Medical Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: July 2009 to August 2013
Groups:
- RAD001 Group: RAD001 will be administered orally as once daily dose of 10 mg (one 10mg tablet or two 5mg tablets) continuously from study day 1 until progression of disease or unacceptable toxicity.
  RAD001: Taken orally once a day in the morning
Period: Overall Study
Arm/Group | RAD001 Group
Started | 50
Participants With Medullary Thyroid Cancer | 10
Completed | 0
Not Completed | 50
Not completed — Death | 3
Not completed — Progression | 29
Not completed — Withdrawal by Subject | 5
Not completed — Adverse Event | 1
Not completed — Physician Decision | 7
Not completed — Still on protocol treatment/ No documentation to say off protocol treatment | 4
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm A: RAD001 will be administered orally as once daily dose of 10 mg (one 10mg tablet or two 5mg tablets) continuously from study day 1 until progression of disease or unacceptable toxicity.
  RAD001: Taken orally once a day in the morning
Arm/Group | Arm A
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 63 [26 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 42
  More than one race | 3
  Unknown or Not Reported | 0
Subtype [Count of Participants; unit: Participants]
  Medullary | 10
  Differentiated | 33
  Anaplastic | 7
Previous Therapies [Count of Participants; unit: Participants]
  Tyrosine Kinase Inhibitors: Yes | 22
  Tyrosine Kinase Inhibitors: No | 28
  Surgery: Yes | 44
  Surgery: No | 6
  Radioactive Iodine: Yes | 31
  Radioactive Iodine: No | 19
  External Beam Radiotherapy: Yes | 30
  External Beam Radiotherapy: No | 20
ECOG Performance Status [Count of Participants; unit: Participants]
  0 - Fully Active | 32
  1 - Restricted | 14
  2- Ambulatory and Capable of Self Care | 4
Site of Distant Metastasis [Count of Participants; unit: Participants]
  None: Yes | 1
  None: No (Not a Metastatic Site) | 49
  Bone: Yes | 21
  Bone: No (Not a Metastatic Site) | 29
  Lung: Yes | 33
  Lung: No (Not a Metastatic Site) | 17
  Liver: Yes | 14
  Liver: No (Not a Metastatic Site) | 36
  Lymph Nodes: Yes | 26
  Lymph Nodes: No (Not a Metastatic Site) | 24
  Other: Yes | 12
  Other: No (Not a Metastatic Site) | 38

OUTCOME MEASURES:

1. Primary Outcome: Median Progression Free Survival
Description: Progression free survival (PFS) is defined as the time from start of treatment to disease progression or death from any cause as estimated by Kaplan Meier methods. Progression is measured using RECIST 1.1 criteria, defined as at least a 20% increase in size in target lesion and/or unequivocal progression of non-target lesions and/or appearance of new lesions. Patients who have not progressed and are alive are censored at the date the patient is known to be progression-free.
Time Frame: Every 2 months for first 24 months, then every 3 months from >24 to 60 months; up to 48 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A
Number analyzed (Participants) | 50
months | 12.5 [7.2 to 17.5]
Statistical Analysis 1: Comparison: Arm A; We will declare the trial a success after observing 7 or more patients with PFS within 6 months. The study will have alpha = 0.092 and power =0.970, assuming a 6 month PFS probability of 0.12 for the null and a PFS probability of 0.35 as the alternative hypothesis; Test type: Other; 6 month PFS probability = 0.35

2. Secondary Outcome: Objective Response Rate
Description: The objective response rate is the proportion of participants achieving complete response (CR) or partial response (PR) on treatment based on Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1) criteria.
  PR or better is achieved if the following are true:
  Target Lesions:
  -At least a 30% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
  Non-target Lesions:
  No progression. No appearance new lesions or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
  Bone Lesions:
  ->50% increase in lesions.
  -No new lesions.
Time Frame: Every 2 months for first 24 months, then every 3 months from >24 to 60 months; up to 48 months.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A
Number analyzed (Participants) | 50
percentage of participants | 6 [0 to 12.6]

3. Secondary Outcome: Median Overall Survival
Description: Overall Survival (OS) is defined as the time from randomization (or registration) to death due to any cause, or censored at date last known alive.
Time Frame: Every 2 months for first 24 months, then every 3 months from >24 to 60 months; up to 5 years post study registration.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A
Number analyzed (Participants) | 50
months | 32.7 [18.7 to 61.3]

4. Secondary Outcome: Mean Change in Quality of Life [Medullary Thyroid Cancer Population Only]
Description: The M. D. Anderson Symptom Inventory (MDASI) questionnaire was used to assess quality of life. Questions 1 to 19 were scored. Each of the 19 questions have a response range of 0 - 10, where 0 represents "not present" and 10 represents "as bad as you can imagine". The 19 responses are averaged together to create a mean score, with a lower score indicating a better quality of life. All questionnaire mean scores at each timepoint are averaged together to give a mean score at that timepoint (baseline and week 8) The mean change in quality of life is calculated by subtracting the baseline mean score from the week 8 mean score.
Time Frame: Measured at baseline and then again at cycle 8 (8 months).
Population: Only 8 of the 10 participants with Medullary Thyroid Cancer filled out both questionnaires (one at baseline and one at cycle 8).
Measure: Mean (Standard Deviation); unit: mean change in score on the MDASI scale
Groups:
- Arm A: RAD001 will be administered orally as once daily dose of 10 mg (one 10mg tablet or two 5mg tablets) continuously from study day 1 until progression of disease or unacceptable toxicity.
  RAD001
Arm/Group | Arm A
Number analyzed (Participants) | 8
mean change in score on the MDASI scale | -0.0621 (0.992)

ADVERSE EVENTS:
Time Frame: Assessed while on treatment and then up to 30 days after discontinuing treatment; up to 31 months
Arm/Group | Arm A
All-Cause Mortality (participants affected / at risk) | 3/50
Serious Adverse Events (participants affected / at risk) | 36/50
Other Adverse Events (participants affected / at risk) | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=50)
Hemoglobin (Blood and lymphatic system disorders) | 3
Hematologic-other (Blood and lymphatic system disorders) | 1
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 1
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 5
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 2
GI-other (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 7
Fever w/o neutropenia (General disorders) | 1
Constitutional, other (General disorders) | 1
Infection w/ gr3-4 neut, skin (Infections and infestations) | 1
Infection Gr0-2 neut, lung (Infections and infestations) | 1
Infection Gr0-2 neut, pharynx (Infections and infestations) | 1
Infection Gr0-2 neut, upper airway (Infections and infestations) | 1
Infection-other (Infections and infestations) | 6
Lymphopenia (Investigations) | 2
Neutrophils (Investigations) | 4
Platelets (Investigations) | 3
Weight loss (Investigations) | 5
ALT, SGPT (Investigations) | 1
Amylase (Investigations) | 2
Hypercholesterolemia (Investigations) | 3
Creatinine (Investigations) | 1
Lipase (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 4
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 1
Joint, pain (Musculoskeletal and connective tissue disorders) | 1
Taste disturbance (Nervous system disorders) | 2
Neurologic-other (Nervous system disorders) | 1
Head/headache (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=50)
Cardiac-ischemia (Cardiac disorders) | 1
Pericardial effusion (non-malignant) (Cardiac disorders) | 2
Tootheache (Gastrointestinal disorders) | 1
Dysgeunsia (Nervous system disorders) | 1
Vascular Disorder - Other (Vascular disorders) | 1
Infection Gr0-2 neut, upper airway (Infections and infestations) | 2
Infection w/ unk ANC lung (Infections and infestations) | 1
Infection w/ unk ANC upper airway NOS (Infections and infestations) | 1
Infection w/ unk ANC urinary tract NOS (Infections and infestations) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Speech impairment (Nervous system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 28
Hemolysis (Blood and lymphatic system disorders) | 1
Hematologic-other (Blood and lymphatic system disorders) | 7
Lymphatics-other (Blood and lymphatic system disorders) | 3
Sinus tachycardia (Cardiac disorders) | 2
Arrhythmia-other (Cardiac disorders) | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Middle ear, pain (Ear and labyrinth disorders) | 1
Dry eye syndrome (Eye disorders) | 1
Ocular surface disease (Eye disorders) | 1
Vision-blurred (Eye disorders) | 1
Vision-photophobia (Eye disorders) | 1
Tearing (Eye disorders) | 1
Ocular-other (Eye disorders) | 3
Chelitis (Gastrointestinal disorders) | 1
Ascites (non-malignant) (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 27
Distention/bloating, abdominal (Gastrointestinal disorders) | 5
Dry mouth (Gastrointestinal disorders) | 17
Dysphagia (Gastrointestinal disorders) | 7
Flatulence (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 6
Hemorrhoids (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Incontinence, anal (Gastrointestinal disorders) | 2
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 25
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 13
Salivary (Gastrointestinal disorders) | 1
Ulcer, gastric (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 11
GI-other (Gastrointestinal disorders) | 12
Anus, hemorrhage (Gastrointestinal disorders) | 1
Oral cavity, hemorrhage (Gastrointestinal disorders) | 2
Rectum, hemorrhage (Gastrointestinal disorders) | 1
Abdomen, pain (Gastrointestinal disorders) | 5
Dental/teeth/peridontal, pain (Gastrointestinal disorders) | 2
Oral cavity, pain (Gastrointestinal disorders) | 2
Oral gums, pain (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 40
Fever w/o neutropenia (General disorders) | 11
Constitutional, other (General disorders) | 3
Edema head and neck (General disorders) | 4
Edema limb (General disorders) | 22
Chest/thoracic pain NOS (General disorders) | 4
Face, pain (General disorders) | 1
Pain NOS (General disorders) | 1
Pain-other (General disorders) | 19
Flu-like syndrome (General disorders) | 1
Syndromes-other (General disorders) | 1
Hepatic-other (Hepatobiliary disorders) | 1
Liver, pain (Hepatobiliary disorders) | 2
Allergic reaction (Immune system disorders) | 2
Allergy-other (Immune system disorders) | 3
Infection w/ gr3-4 neut, lung (Infections and infestations) | 1
Infection Gr0-2 neut, dental-tooth (Infections and infestations) | 1
Infection Gr0-2 neut, eye NOS (Infections and infestations) | 1
Infection Gr0-2 neut, lung (Infections and infestations) | 2
Infection Gr0-2 neut, middle ear (Infections and infestations) | 1
Infection Gr0-2 neut, oral cavity (Infections and infestations) | 1
Infection Gr0-2 neut, salivary (Infections and infestations) | 1
Infection Gr0-2 neut, sinus (Infections and infestations) | 1
Infection Gr0-2 neut, skin (Infections and infestations) | 1
Infection Gr0-2 neut, ungual (Infections and infestations) | 1
Infection Gr0-2 neut, urinary tract (Infections and infestations) | 3
Infection w/ unk ANC sinus (Infections and infestations) | 1
Infection-other (Infections and infestations) | 17
Wound - non-infectious (Injury, poisoning and procedural complications) | 2
Leukocytes (Investigations) | 10
Lymphopenia (Investigations) | 7
Neutrophils (Investigations) | 9
Platelets (Investigations) | 13
Weight gain (Investigations) | 3
Weight loss (Investigations) | 21
Coagulation-other (Investigations) | 1
Alkaline phosphatase (Investigations) | 6
ALT, SGPT (Investigations) | 13
Amylase (Investigations) | 2
AST, SGOT (Investigations) | 18
Hypercholesterolemia (Investigations) | 29
Creatinine (Investigations) | 7
Lipase (Investigations) | 1
Metabolic/Laboratory-other (Investigations) | 3
Pancreatic glucose intolerance (Metabolism and nutrition disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 24
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Alkalosis (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 12
Hyperglycemia (Metabolism and nutrition disorders) | 16
Hypoglycemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 8
Hypernatremia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 4
Hypertriglyceridemia (Metabolism and nutrition disorders) | 19
Nonneuropathic lower extr muscle weak (Musculoskeletal and connective tissue disorders) | 2
Nonneuropathic upper extr muscle weak (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 4
Back, pain (Musculoskeletal and connective tissue disorders) | 17
Bone, pain (Musculoskeletal and connective tissue disorders) | 5
Chest wall, pain (Musculoskeletal and connective tissue disorders) | 4
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 10
Joint, pain (Musculoskeletal and connective tissue disorders) | 11
Muscle, pain (Musculoskeletal and connective tissue disorders) | 3
Neck, pain (Musculoskeletal and connective tissue disorders) | 4
Taste disturbance (Nervous system disorders) | 19
Dizziness (Nervous system disorders) | 9
Neuropathy CN VIII hearing + balance (Nervous system disorders) | 1
Neuropathy-motor (Nervous system disorders) | 1
Neuropathy-sensory (Nervous system disorders) | 4
Tremor (Nervous system disorders) | 2
Neurologic-other (Nervous system disorders) | 1
Head/headache (Nervous system disorders) | 15
Neuropathic, pain (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 16
Confusion (Psychiatric disorders) | 3
Anxiety (Psychiatric disorders) | 9
Depression (Psychiatric disorders) | 5
Libido (Psychiatric disorders) | 1
Urinary hemorrhage NOS (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Bladder, pain (Renal and urinary disorders) | 1
Urethra, pain (Renal and urinary disorders) | 1
Cystitis (Renal and urinary disorders) | 1
Incontinence urinary (Renal and urinary disorders) | 1
Obstruction-bladder (Renal and urinary disorders) | 1
Obstruction-ureteral (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 5
Urine color (Renal and urinary disorders) | 1
Renal/GU-other (Renal and urinary disorders) | 2
Pelvic, pain (Reproductive system and breast disorders) | 2
Scrotum, pain (Reproductive system and breast disorders) | 1
Testicle, pain (Reproductive system and breast disorders) | 1
Sexual/Reproductive function-Other (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 8
Pleura, pain (Respiratory, thoracic and mediastinal disorders) | 1
Throat/pharynx/larynx, pain (Respiratory, thoracic and mediastinal disorders) | 7
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 31
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 28
Edema, larynx (Respiratory, thoracic and mediastinal disorders) | 1
Fistula trachea (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 5
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 5
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 7
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 8
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 12
Sweating (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 8
Alopecia (Skin and subcutaneous tissue disorders) | 2
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Induration/fibrosis (Skin and subcutaneous tissue disorders) | 1
Nail changes (Skin and subcutaneous tissue disorders) | 8
Pruritus/itching (Skin and subcutaneous tissue disorders) | 4
Rash/desquamation (Skin and subcutaneous tissue disorders) | 5
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 22
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 1
Ulceration (Skin and subcutaneous tissue disorders) | 1
Skin-other (Skin and subcutaneous tissue disorders) | 16
Skin, pain (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 7
Hypotension (Vascular disorders) | 1
Flushing (Vascular disorders) | 1
Hot flashes (Vascular disorders) | 1
Hemorrhage-other (Vascular disorders) | 2
Dermal change lymphedema (Vascular disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 3
Vascular-Other (Specify) (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-28): https://cdn.clinicaltrials.gov/large-docs/58/NCT00936858/Prot_SAP_000.pdf